CLINICAL TRIAL: NCT02625636
Title: A Randomized, Double-blind, Glucagon and Placebo-controlled Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Single Escalating Doses of SAR438544 Administered by Subcutaneous Route in Healthy Subjects and Patients With Type 1diabetes Mellitus
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of Escalating Doses of SAR438544 in Comparison to Placebo and Glucagon in Healthy Subjects and Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TDU14518; U1111-1172-1152 (Other: UTN)
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SAR438544 dose 1 (Experimental): Single dose of SAR438544 given SC under fasting conditions
  Interventions: Drug: SAR438544
- SAR438544 dose 2 (Experimental): Single dose of SAR438544 given SC under fasting conditions
  Interventions: Drug: SAR438544
- SAR438544 dose 3 (Experimental): Single dose of SAR438544 given SC under fasting conditions
  Interventions: Drug: SAR438544
- Placebo (Placebo Comparator): Single dose of placebo given SC under fasting conditions
  Interventions: Drug: placebo
- Glucagon (Active Comparator): Single dose of glucagon given SC under fasting conditions
  Interventions: Drug: r-glucagon
- SAR438544 Optional Dose (Experimental): Optional lower, intermediate, or higher dose of SAR438544 given SC under fasting conditions
  Interventions: Drug: SAR438544

INTERVENTIONS:
Drug: SAR438544 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: SAR438544 Optional Dose; SAR438544 dose 1; SAR438544 dose 2; SAR438544 dose 3
Drug: placebo — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Placebo
Drug: r-glucagon — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: GlucaGen® HypoKit, glucagon
  Arms: Glucagon

SUMMARY:
Primary Objective:

To assess the tolerability and safety of SAR438544 after single ascending subcutaneous (SC) doses in healthy subjects and in type 1 diabetes mellitus (T1DM) patients.

Secondary Objective:

To assess the preliminary pharmacodynamics (PD) and pharmacokinetic (PK) parameters of SAR438544 after single ascending SC doses in healthy subjects and in T1DM patients.

DETAILED DESCRIPTION:
Healthy subjects:

The total duration of study per subject is up to 4.5 weeks with 2 to 21 days screening period, 1 day for treatment, and 7 days (+/- 1 day) follow-up after IMP administration.

T1DM patients:

The total duration of study per patient is up to 5.5 weeks with 3 to 28 days screening period, 1 day for treatment, and 7 days (+/- 1 day) follow-up after IMP administration.

One or more interim analyses may be performed to support decisions for the next steps of the study.

ELIGIBILITY:
Inclusion criteria :

Healthy subjects:

* Male or female subjects, between 18 and 45 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Female subject must use a double contraception method, including a highly effective method of birth control, except if she has undergone sterilization defined as tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and bilateral tubal ligation at least 3 months earlier or is postmenopausal.
* The accepted double contraception methods include the use of intrauterine device or hormonal contraception started at least 30 days prior to the screening start and continued for at least 3 months after IMP dosing in addition to one of the following contraceptive options: (1) condom plus spermicide; (2) diaphragm plus spermicide or cervical/vault cap plus spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma FSH level >30 UI/L in women older than 40 years of age
* Having given written informed consent prior to undertaking any study-related procedure.
* Not under any administrative or legal supervision.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom, diaphragm or cervical cap, plus spermicide) plus (intra-uterine device or hormonal contraceptive) from the inclusion up to 3 months after the last dosing (except if sterilized).
* Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 3 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 3 months after the last dosing.

T1DM patients:

* Male or female patients, between 18 and 60 years of age, inclusive, with T1DM for at least one year, as defined by the American Diabetes Association.
* Total (basal+short acting) daily insulin dose of <1.2 U/kg/day.
* Body weight between 50.0 and 110 kg, inclusive, the BMI between 18.5 and 30.0 kg/m^2, inclusive.
* Fasting serum C-peptide <0.3 nmol/L.
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9%).
* Stable insulin regimen for at least 2 months prior to study and self-monitoring of blood glucose before screening visit.
* Certified as otherwise healthy for T1DM by assessment of medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculoskeletal system), unless the Investigator considers any abnormality to be clinically irrelevant and not interfering with the conduct of the study.
* Female subject must use a double contraception method, including a highly effective method of birth control, except if she has undergone sterilization defined as tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and bilateral tubal ligation at least 3 months earlier or is postmenopausal.
* The accepted double contraception methods include the use of intrauterine device or hormonal contraception started at least 30 days prior to the screening start and continued for at least 3 months after IMP dosing in addition to one of the following contraceptive options: (1) condom plus spermicide; (2) diaphragm plus spermicide or cervical/vault cap plus spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma FSH level >30 UI/L in women older than 40 years of age.
* Having given written informed consent prior to undertaking any study-related procedure.
* Not under any administrative or legal supervision.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom, diaphragm or cervical cap, plus spermicide) plus (intra-uterine device or hormonal contraceptive) from the inclusion up to 3 months after the last dosing (except if sterilized).
* Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 3 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 3 months after the last dosing.

Exclusion criteria:

Healthy subjects:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of any drug allergy or allergic disease that in the opinion of the Investigator may interfere with subject safety or data integrity during the study.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-HCG] blood test), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or PD half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab) and human immunodeficiency virus 1 antigen (HIV1 Ag).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol breath test.

T1DM patients:

* Any history or presence of clinically relevant cardiovascular (includes ischemia, atrioventricular [AV] block; arrhythmias), pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent severe headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood loss (>300 mL) within 3 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of any drug allergy or allergic disease that in the opinion of the Investigator may interfere with patient safety or data integrity during the study.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* If female, pregnancy (defined as positive β-HCG blood test), breast-feeding at screening and before any treatment periods (defined as positive β-HCG urine test).
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Positive result on any of the following tests: HBs Ag, anti-HCV Abs, anti-HIV1 and anti-HIV2 Abs and HIV1 Ag.
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol breath test.
* Known hypersensitivity to glucagon, lactose or any other constituent in GlucaGen^® HypoKit and SAR438544 and their excipients.
* Any contraindication from the use of glucagon:
* Pheochromocytoma
* Insulinoma and glucagonoma

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Day 1 to Day 7 (+/- 1 day)

SECONDARY OUTCOMES:
Assessment of PD parameter: continuous monitoring of blood glucose levels over a period of 6 hours post-dose | Day 1
Assessment of PD parameter: area under plasma concentration of the BG-time curve between investigational medicinal product (IMP) dosing and time t (BG-AUC0-t) | Day 1
Assessment of PD parameter: BG-maximum concentration (BG-Cmax) | Day 1
Assessment of PD parameter: BG-time to Cmax (BG-tmax) | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): Cmax | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): tmax | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): tlast | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): terminal half life | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): area under curve from zero time until the last measurable concentration (AUClast) | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): AUC | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): partial AUCs (AUC0-t) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Chula Vista, California, United States